CLINICAL TRIAL: NCT03774914
Title: International LEMTRADA Pregnancy Exposure Cohort in Multiple Sclerosis
Brief Title: LEMTRADA Pregnancy Registry in Multiple Sclerosis
Status: Terminated | Type: Observational
Why Stopped: The sponsor stopped the study due to low recruitment with no safety concerns
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: OBS13436; EU PAS - cat 3
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04-21

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lemtrada: Pregnant women exposed to LEMTRADA which is administered by IV infusion for 5 consecutive days, then for 3 consecutive days, 12 months after the first/previous treatment course
  Interventions: Drug: Alemtuzumab (GZ402673)

INTERVENTIONS:
Drug: Alemtuzumab (GZ402673) — Pharmaceutical form:Concentrate for solution for infusion Route of administration: Intravenous infusion
  Other Names: Lemtrada

SUMMARY:
Primary Objective:

The primary goal of this registry is to assess the risk of spontaneous abortion in prospective enrolled women exposed to LEMTRADA for multiple sclerosis.

Secondary Objective:

The secondary goals of this registry is to assess maternal, fetal and infant outcome in women with multiple sclerosis, exposed to LEMTRADA.

DETAILED DESCRIPTION:
From enrollment during pregnancy up to 1 year after delivery for infant follow-up (maximum approximatively 20 months)

ELIGIBILITY:
Inclusion criteria :

* Women with Multiple Sclerosis who were or became pregnant within the period of time between the first infusion of a course of treatment with LEMTRADA to 4 months after their last infusion for that course.
* Women able and willing to provide informed consent for study participation and the requirement of the study. Informed consent will be obtained at the time of enrollment in accordance with local regulatory requirements.

Exclusion criteria:

- Previous enrollment in this study for a previous pregnancy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with Multiple Sclerosis who were or became pregnant within the period of time between the first infusion of a course of treatment with LEMTRADA to 4 months after their last infusion for that course.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Spontaneous abortions (≤20 weeks gestation) | 32 weeks gestation
  Number and rate of spontaneous abortions on pregnant women prospectively enrolled (pregnancy outcome unknown at time of enrollment)

SECONDARY OUTCOMES:
Major congenital malformations | From birth to 1 year after delivery
  Numbers and rates of major congenital malformations on pregnant women prospectively enrolled (pregnancy outcome unknown at time of enrollment)
Minor congenital malformations | From birth to 1 year after delivery
  Numbers and rates of minor congenital malformations on pregnant women prospectively enrolled (pregnancy outcome unknown at time of enrollment)
Stillbirth (any non-deliberate foetal death at >20 weeks gestation) | 26-32 weeks' gestation to within 6 weeks after the end of the pregnancy
  Numbers and rates of stillbirth, on pregnant women prospectively enrolled (pregnancy outcome unknown at time of enrollment)
Full-term live birth i.e. infants born maturely (≥37 gestation weeks) | Within 6 weeks after the end of the pregnancy
  Numbers and rates of full-term live birth on pregnant women prospectively enrolled (pregnancy outcome unknown at time of enrollment)
Preterm birth i.e. infants born prematurely i.e., live-born infant i.e., (pre-term <37 weeks) | 26-32 weeks' gestation to within 6 weeks after the end of the pregnancy
  Numbers and rates of pre-term birth on pregnant women prospectively enrolled (pregnancy outcome unknown at time of enrollment)
Elective terminations i.e. any induced or voluntary fetal loss | 16-20 weeks' gestation
  Numbers and rates of elective terminations on pregnant women prospectively enrolled (pregnancy outcome unknown at time of enrollment)
Small for gestational age at birth i.e. birth size (weight, length, or head circumference) ≤10th percentile for gender and gestational age | Within 6 weeks after the end of the pregnancy
  Numbers and rates of small for gestational age on pregnant women prospectively enrolled (pregnancy outcome unknown at time of enrollment)
Any other adverse pregnancy outcomes | Baseline to week 40
  Numbers of adverse events
Infant postnatal growth (up to the first year of life) | 1 year after delivery
  Numbers and rates of infants with postnatal size (weight, length or head circumference) less than or equal to the 10th percentile for sex and age using National Center for Health Statistics (NCHS) pediatric growth curves, and adjusted postnatal age for premature infants.
Infant development impairment (up to the first year of life) | 1 year after delivery
  Numbers and rates of infants with development impairment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- Investigational Site Number :840999, New York, New York, United States
- Investigational Site Number :036001, Box Hill, Victoria, Australia
- Investigational Site Number :040-001, Linz, Austria
- Investigational Site Number :56, Charleroi, Belgium
- Investigational Site Number :124999, Canada, Canada
- Investigational Site Number :208001, Aarhus C, Denmark
- Investigational Site Number :276001, Bochum, Germany
- Investigational Site Number :380001, Gallarate (VA), Italy
- Investigational Site Number :528999, Netherlands, Netherlands
- Investigational Site Number :724999, Spain, Spain
- Investigational Site Number :752001, Gothenburg, Sweden
- Investigational Site Number :756001, Zurich, Switzerland
- Investigational Site Number :826-001, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org